CLINICAL TRIAL: NCT05397847
Title: The Effect of Nursing Interventions Applied at Home for Rational Drug Use and Raising Awareness in Elderly Individuals
Brief Title: Rational Drug Use in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, BUSRA ALTINEL, Dr, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 555444
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Rational Drug Use
Keywords: rational drug use; elderly individuals; nurse; education
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Education, rational drug use guide and consultancy services will be provided to elderly individuals through home visits.
  Interventions: Behavioral: Education; Other: Rational Drug Use Guide; Other: Medicine Box; Behavioral: Counseling
- Control (No Intervention): No intervention will be made to the control group, and after the post-test, the rational drug use guide and the medicine box will also be given to the control group.

INTERVENTIONS:
Behavioral: Education — Rational Drug Use in Elderly Individuals
  1. Training: Through home visits, an average of 30 minutes of training will be given to elderly individuals (drugs, rational drug use, the importance of rational drug use, and what the elderly should do for rational drug use). Question-answer method and visual materials will be used in the training.
  2. Training: An average of 20 minutes of training will be given, including a brief repetition of the topics covered in the first training, via a home visit. Visual materials will be used in the training.
  Arms: Experiment
Other: Rational Drug Use Guide — At the end of the first training, a rational drug use guide will be given to elderly individuals, including the topics explained.
  Arms: Experiment
Other: Medicine Box — Elderly individuals will be given a medicine box large enough to be carried in the pocket when appropriate, so that the elderly people do not forget their medicines and use them regularly, with a 7-day medicine compartment that organizes their medicines and a daily (morning, noon, evening and night) medicine box.
  Arms: Experiment
Behavioral: Counseling — After the training, counseling services will be given to elderly individuals regarding rational drug use. Within the scope of the counseling service, it will be ensured that the drugs used by the elderly person are regulated and their questions about rational drug use will be answered.
  Arms: Experiment

SUMMARY:
Irrational drug use, which is an important public health problem worldwide, is common in the elderly. While irrational drug use negatively affects all age groups, it poses a significant threat to the health of the elderly. This study aims to examine the effects of 8-week interventions, which include training, counseling and awareness-raising nursing practices for rational drug use and awareness development, through home visits to elderly individuals; planned in a randomized controlled experimental design.

The research will be carried out between May-July 2022 in Halkapınar Central Family Health Center located in Konya province Halkapınar district. The study group will be randomly assigned 35 experimental and 35 control groups, a total of 70 elderly individuals. Attempts made for the experimental group for eight weeks; Education through home visits on rational drug use will include counseling, guidance on rational drug use, and the delivery of a medicine box. The control group will continue with the routine applications. Taking into account the right of the control group to be informed about ethics after the post-tests, the training, guide and medicine box will also be given to the control group through home visits given to the experimental group. Data will be collected by face-to-face interview method using the Elderly Information Form, Rational Drug Use Scale and Rational Drug Use Awareness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Be 65 years or older
* Living in Halkapınar
* Registering with the Central Family Health Centre
* Be able to speak Turkish

Exclusion Criteria:

* Having a score below 24 on the Standardized Mini Mental Test
* Having any communication or medically diagnosed mental problems
* Being bedridden
* Having a neurological problem

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Using medicine with care | 6 weeks
  Rational drug use scale mean scores of elderly individuals
Rational Drug Use Awareness | 6 weeks
  Rational Drug Use Awareness Scale mean scores of elderly individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes